CLINICAL TRIAL: NCT05938738
Title: A Portable Dyspnea Relief Device for Episodic Breathlessness in COPD (PEP-buddy): Effect on Dyspnea Severity and Mechanism of Action
Brief Title: PEP-buddy in COPD: Effect on Dyspnea Severity and Mechanism of Action
Acronym: RELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JE Hartman, Principal investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RELIEF
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEP-buddy (Experimental): Patients will use the PEP-buddy as needed.
  Interventions: Device: PEP-buddy

INTERVENTIONS:
Device: PEP-buddy — PEP-buddy

SUMMARY:
Chronic dyspnea is the most characteristic symptom of patients with Chronic Obstructive Pulmonary Disease (COPD), with intermittent increases during exercise and other events.Despite optimal standard therapy, episodic dyspnea is a common occurrence in COPD. Recently, the PEP buddy was developed which is an easy-to use, hands-free device that generates positive expiratory pressure (PEP). Although currently the available evidence is limited, it indicates that utilizing the PEP-buddy can result in enhancements in dyspnea during exertion, exertional desaturation and overall quality of life. More research is needed to evaluate the effectiveness of this device and the long term usability, as well as getting more insight in the mechanism of action. Therefore, the aim of our study is to explore the potential of this device for patients with COPD and episodic breathlessness.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years
2. Read, understood and signed Informed Consent
3. COPD Gold class II-IV/ B or E (FEV1<60% of predicted, CAT ≥10 points)

5. Optimized standard therapy according to the study physician 6. Episodic breathlessness requiring intervention (i.e. taking rest during physical activities, as needed inhalation medication, breathing techniques, as needed opioids) at least three days per week

Exclusion Criteria:

1. Other severe disease causing episodic breathlessness
2. Life expectancy ≤ 3 months
3. Exacerbation of COPD 4 weeks prior to inclusion
4. Change in COPD management targeted at breathlessness 8 weeks prior to inclusion
5. Inability to use the PEP buddy device
6. Currently participating in another interventional clinical study
7. Any other conditions, which, in the opinion of the investigator would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dyspnea severity | 4 weeks
  To investigate the effect of the portable dyspnea relief device on dyspnea severity after 4 weeks. Dyspnea severity is measured by the dyspnea domain of the chronic respiratory questionnaire (CRQ), this score of this scale ranges from 5-35, with a higher score indicating more severe dyspnea.

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No